CLINICAL TRIAL: NCT00629980
Title: A Multi-Center, Open-Label, Randomized Pilot Study of the Safety and Efficacy of AzaSite® Ophthalmic Solution, 1% in Combination With Mechanical Therapy Versus Mechanical Therapy Alone in Subjects With Blepharitis
Brief Title: Safety and Efficacy Pilot Study of AzaSite® (Azithromycin) in Subjects With Blepharitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Mike Schiewe, Inspire Pharmaceuticals, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 041-105; P08651
Record Dates: First submitted 2008-02-27; First posted 2008-03-06 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Blepharitis
MeSH Terms: conditions — Blepharitis | interventions — Azithromycin

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AzaSite®
- 2 (No Intervention)

INTERVENTIONS:
Drug: AzaSite® — ophthalmic solution; 1 drop in each eye BID for two days, then 1 drop in each eye QD for ~26 days
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of AzaSite® ophthalmic solution, 1% on signs and symptoms of blepharitis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of moderate to severe chronic blepharitis
* if female of childbearing potential, are non-pregnant and non-lactating

Exclusion Criteria:

* had ocular surface surgery (LASIK, refractive, etc.) within the past year
* unwilling to discontinue the use of contact lenses during the study
* have glaucoma
* unable or unwilling to withhold the use of lid scrubs during the study
* have a serious systemic disease or uncontrolled medical condition that in the judgment of the investigator could confound study assessments or limit compliance
* currently using any preserved topical ocular medications (with the exception of unpreserved tear substitutes) at the time of entry into the study or during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
change in clinical signs and symptoms associated with blepharitis | 4 weeks

SECONDARY OUTCOMES:
standard ocular safety assessments | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Reza Haque, MD, Study Director — Sponsor GmbH
Locations (9):
- United States (9):
  - Sall Research Medical Center, Artesia, California
  - North Valley Eye Medical Group, Mission Hills, California
  - Center for Excellence in Eye Care, Miami, Florida
  - Kentuckiana Institute for Eye Research, Louisville, Kentucky
  - Tauber Eye Center, Kansas City, Missouri
  - Silverstein Eye Centers, Kansas City, Missouri
  - South Shore Eye Care, LLP, Wantagh, New York
  - Toyos Clinic, Jackson, Tennessee
  - Corona Research Consultants, Inc., El Paso, Texas